CLINICAL TRIAL: NCT06654323
Title: The Dose Trial: Dose Intensity of Behavioral Interventions for Childhood Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Bill Heerman, Assoc Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 241527; BPS-2023C1-31064 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2024-10-02; First posted 2024-10-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Childhood Obesity
Keywords: Behavioral Intervention; Rural and Urban Populations; Racial and Ethnic Minority Populations; Nutrition Counseling; Community Resource Counseling
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 26-hour intensive behavioral lifestyle intervention (Experimental): Participants will receive 4 visits, (1 hour total) with their child's pediatric primary care provider, on-demand web-based learning modules that focus on building skills and knowledge in health behaviors (7 hours), community resource counseling sessions delivered by a social worker or similar healthcare professional (4 sessions, 2 hours total), and personalized nutrition counseling delivered by a registered dietitian or similar healthcare professional: 16 sessions (60 minutes per session).
  Interventions: Behavioral: Intensive Behavioral Lifestyle Modification
- 22-hour intensive behavioral lifestyle intervention (Active Comparator): Participants will receive 4 visits, (1 hour total) with their child's pediatric primary care provider, on-demand web-based learning modules that focus on building skills and knowledge in health behaviors (7 hours), community resource counseling sessions delivered by a social worker or similar healthcare professional (4 sessions, 2 hours total), and personalized nutrition counseling delivered by a registered dietitian or similar healthcare professional for 12 sessions (60 minutes per session).
  Interventions: Behavioral: Intensive Behavioral Lifestyle Modification
- 19-hour intensive behavioral lifestyle intervention (Active Comparator): Participants will receive 4 visits, (1 hour total) with their child's pediatric primary care provider, on-demand web-based learning modules that focus on building skills and knowledge in health behaviors (7 hours), community resource counseling sessions delivered by a social worker or similar healthcare professional (4 sessions, 2 hours total), and personalized nutrition counseling delivered by a registered dietitian or similar healthcare professiona for 9 sessions (60 minutes per session).
  Interventions: Behavioral: Intensive Behavioral Lifestyle Modification
- 16-hour intensive behavioral lifestyle intervention (Active Comparator): Participants will receive 4 visits, (1 hour total) with their child's pediatric primary care provider, on-demand web-based learning modules that focus on building skills and knowledge in health behaviors (7 hours), community resource counseling sessions delivered by a social worker or similar healthcare professional (4 sessions, 2 hours total), and personalized nutrition counseling delivered by a registered dietitian or similar healthcare professional for 8 sessions (45 minutes per session).
  Interventions: Behavioral: Intensive Behavioral Lifestyle Modification
- 13-hour intensive behavioral lifestyle intervention (Active Comparator): Participants will receive 4 visits, (1 hour total) with their child's pediatric primary care provider, on-demand web-based learning modules that focus on building skills and knowledge in health behaviors (7 hours), community resource counseling sessions delivered by a social worker or similar healthcare professional (4 sessions, 2 hours total), and personalized nutrition counseling delivered by a registered dietitian or similar healthcare professional for 6 sessions (30 minutes per session).
  Interventions: Behavioral: Intensive Behavioral Lifestyle Modification

INTERVENTIONS:
Behavioral: Intensive Behavioral Lifestyle Modification — Participants in all arms will receive visits with their child's primary care provider (4 visits, 1 hour total), on-demand web-based learning modules that focus on building skills and knowledge in health behaviors (7 hours), and community resource counseling sessions delivered by a social worker or similar healthcare professional (4 sessions, 2 hours total). The difference between arms will be in the frequency and duration of personalized nutrition counseling delivered by a registered dietitian or similar healthcare professional: 16 sessions (60 minutes per session), 12 sessions (60 minutes per session), 9 sessions (60 minutes per session), 8 sessions (45 minutes per session), or 6 sessions (30 minutes per session).

SUMMARY:
The research team is recruiting 900 children between the ages 5-17 with obesity from Tennessee and Louisiana. The team is assigning children and their caregivers by chance to one of five groups. In the first group, 300 children and their caregivers receive 26 hours of IBT. In the second group, 300 children and their caregivers receive 13 hours of IBT. The remaining three groups of 100 children and their caregivers receive 16, 19, or 22 hours of IBT.

Children's healthcare providers, nutritionists, and social workers are providing IBT to each of the groups over six months. At the start of the study and again after one year, the research team is measuring the children's body mass index, or BMI. BMI is a measure of a person's body fat based on their height and weight. The team is also looking at the children's:

* Diet
* Exercise
* Sleep
* Media use
* Quality of life

DETAILED DESCRIPTION:
The Dose study aims to evaluate the optimal number of contact hours (i.e., dose) of intensive behavioral lifestyle interventions for childhood obesity. Current recommendations by the American Academy of Pediatrics (AAP) and the United States Preventive Services Task Force (USPSTF) suggest that intensive behavioral lifestyle interventions should have at least 26 hours of contact time. This is a difficult standard to achieve, as it requires significant resources from healthcare systems and time from families. This study's purpose is to test whether 26 hours is needed to achieve clinically meaningful reductions in child weight among children with obesity.

The investigators will conduct a randomized clinical trial (RCT) where children are randomized to one of five treatment intensities: 26 hours, 22 hours, 19 hours, 16 hours, or 13 hours. The study will use a non-inferiority design: can equal effectiveness be achieved comparing the 26-hour standard to reduced intensities?

900 children with obesity ages 5-17 years old will be randomized, with a focus on rural and minority communities in Tennessee (TN) and Louisiana (LA). The study will engage approximately 15 clinics in TN and 15 in LA.

The intervention will be integrated into local pediatric primary care practices. Participants in all arms will receive the same number of visits with their child's primary care provider (4 visits, 1 hour total), on-demand web-based learning modules that focus on building skills and knowledge in health behaviors (7 hours), and community resource counseling sessions delivered by a social worker or similar healthcare professional (4 sessions, 2 hours total). The difference between arms will be in the frequency and duration of personalized nutrition counseling delivered by a registered dietitian or similar healthcare professional: 16 sessions (60 minutes per session), 12 sessions (60 minutes per session), 9 sessions (60 minutes per session), 8 sessions (45 minutes per session), or 6 sessions (30 minutes per session).

The primary outcome is child body mass index (BMI) expressed as a percentage of the 95th percentile (%BMIp95) of the CDC growth curves, over 12 months, measured approximately 5 times. Our primary hypothesis is that 13-hours will be non-inferior to 26-hours. The analysis also includes multiple, pre-specified sub-group analyses, as there may be important subgroups who require more than 13 hours (e.g., children with a very high starting BMI). Secondary outcomes include changes in child quality of life and health behaviors. The analysis will assess reach, feasibility, and accessibility of this approach for both participants and pediatric healthcare providers, guided by the RE-AIM framework.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥95th percentile for age and sex based on standardized CDC growth curves.
* parent/caregiver aged ≥ 18 years old
* are comfortable speaking and reading English or Spanish;
* are a patient of a participating clinical practice;
* are able to provide written or verbal consent/assent;
* are able to attend scheduled sessions in the 12-month study;
* are willing to make behavioral and lifestyle changes;
* are able to access the internet to participate in online intervention components;
* complete baseline data collection, including child height and weight; and
* complete at least 90% of baseline survey items no later than 14 days after the baseline visit.

Exclusion Criteria:

* families for whom the primary care provider (PCP) or site principal investigator (PI) thinks the study and/or intervention is clinically/medically inappropriate (e.g. developmental delay, disordered eating, mobility impairments, cognitive or mental difficulties);
* participant child is taking weight management medications at the time of enrollment;
* participant child plans to undergo bariatric surgery or another weight loss operation during the 12-month study; or
* participant caregiver-child dyad has plans to move during the 12-month study and will no longer be a patient of a participating clinic.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Percent of the 95th BMI Percentile | 5 times over 12 months
  The primary outcome is child body mass index (BMI) expressed as a percentage of the 95th percentile (%BMIp95) of the CDC growth curves.

SECONDARY OUTCOMES:
Child Diet | 12 months
  Diet Recall, using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool. A variety of dietary measures will be abstracted from this dietary recall including the total number of calories consumed daily and the Healthy Eating Index (HEI) which has a range of 0-100, where higher numbers represent a healthier diet.
Child physical activity | 12 months
  Physical Activity Questionnaire for Children or Adolescents, which provides a summary physical activity score derived from nine items, each scored on a 5-point scale. High scores represent more physical activity.
Child Media Use | 12 months
  Cumulative Media Use Index, which is a summary score ranging from 0 to 14, where high numbers represent more media use.
Child Sleep | 12 months
  Short Form Children's Sleep Habits Questionnaire, scored with a range of 23 to 39 where a higher score is indicative of more disturbed sleep

CONTACTS AND LOCATIONS:
Overall Officials: William Heerman, MD MPH, Principal Investigator — Vanderbilt University Medical Center; Amanda Staiano, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (2):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No